CLINICAL TRIAL: NCT00450021
Title: Imaging of Cannabinoid CB(1) Receptors Using [11C] MePPEP
Brief Title: Imaging of Cannabinoid Receptors Using New Radioactive Tracer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: National Institute of Mental Health, Eli Lilly & Co. (Unknown)
Responsible Party: Robert B. Innis, M.D./National Institute of Mental Health, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 070118; 07-M-0118
Record Dates: First submitted 2007-03-20; First posted 2007-03-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-02-06

CONDITIONS: Healthy
Keywords: PET; CB1 Receptor; Cannabinoid; [11C] MePPEP; Brain Imaging; Healthy Volunteer; HV
MeSH Terms: interventions — Carbon-11

INTERVENTIONS:
Drug: [(11)C] MePPEP

SUMMARY:
This study will test a new radioactive tracer, [(11)C]MePPEP, for use in positron emission tomography (PET) imaging. The tracer is used to visualize cannabinoid receptors, proteins in the brain that mediate a variety of natural chemicals. These receptors may be important in behavioral diseases such as addiction, obesity and psychiatric diseases.

Healthy normal volunteers between 18 and 65 years of age may be eligible for this study.

Ten participants undergo whole body PET imaging to determine where the [(11)C]MePPEP tracer is distributed in the body in order to calculate radiation exposure from the tracer. Another 10 subjects undergo brain imaging with [(11)C]MePPEP to measure cannabinoid receptors in the brain.

All participants are evaluated with a medical history and physical examination, blood and urine tests and an electrocardiogram (ECG) before scanning. They then have a PET scan. For this procedure, a catheter (plastic tube) is placed in a vein in the arm through which the tracer is injected. A special mask is fitted to the head and attached to the bed to help keep the head in place during the scan. Subjects undergoing brain imaging also have a catheter placed in an artery in the wrist from which blood samples are collected during the procedure. The scan lasts about 2 to 2.5 hours.

Subjects undergoing brain imaging also have magnetic resonance imaging (MRI) within 1 year of the PET scan. For MRI, the subject lies on a bed that moves into the tubular scanner, wearing earplugs to protect the ears from loud noises that occur during the scan. The procedure takes about 1 hour.

DETAILED DESCRIPTION:
BRAIN IMAGING:

OBJECTIVE:

The central cannabinoid receptor, CB(1) is one of the most abundant neuromodulatory receptors in the brain. It is found on glutamatergic, dopaminergic and GABA-ergic synaptic terminals and belongs to the G-protein coupled receptor family. The CB(1) is a target for drug therapy, including the use of an antagonist as an appetite suppressant. The central cannabinoid receptor CB(1) has never been visualized in humans. In collaboration with Eli Lilly, we developed a promising PET ligand for the CB(1) receptor: [(11)C]MePPEP. This study is known by Eli Lilly as H6O-MC-GCEB.

STUDY POPULATION:

In the current protocol, we wish to evaluate [(11)C]MePPEP in approximately 15 healthy subjects.

DESIGN:

Brain imaging studies will consist of subject evaluation followed by PET and MRI scans.

OUTCOME MEASURES:

We intend to determine the kinetics of brain uptake and washout, clearance in the plasma, and the distribution volume of [(11)C]MePPEP calculated with compartmental modeling. Distribution volume is proportional to the density of receptors and is equal to the ratio at equilibrium of uptake in brain to the concentration of parent radiotracer in plasma.

WHOLE BODY DOSIMETRY:

OBJECTIVE:

Should the brain imaging studies prove to be successful, we will continue with whole body dosimetry studies. Preliminary dosimetry studies with [(11)C]MePPEP have been performed in nonhuman primates; however, these need to be continued in humans before further investigation of this novel tracer can continue. This study is known by Eli Lilly as H6O-MC-GCEC.

STUDY POPULATION:

In the current protocol, we wish to evaluate [(11)C]MePPEP in approximately 10 additional healthy subjects.

DESIGN:

The whole body dosimetry studies will consist of subject evaluation followed by a PET scan.

OUTCOME MEASURES:

We intend to determine the whole body distribution of activity and thereby calculate radiation exposure to organs of the body.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must be healthy and aged 18-65 years, with history/physical exam, ECG, and laboratory tests within one year of the PET scan. The volunteer must sign an informed consent form.

EXCLUSION CRITERIA:

1. Current psychiatric illness, substance abuse including marijuana use, or severe systemic disease based on history and physical exam.
2. Laboratory tests with clinically significant abnormalities or positive urine toxicology screen.
3. Prior participation in other research protocols in the last year such that radiation exposure would exceed the annual limits.
4. Pregnancy and breast feeding.
5. Claustrophobia.
6. Presence of ferromagnetic metal in the body or heart pacemaker.
7. Positive HIV test.
8. Employee of the investigative site or an immediate family member of an employee of the investigative site. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
9. Employee of Eli Lilly and Company.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2007-03-19; Primary Completion 2008-02-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of novel PET tracer for DB! in Brain imaging.

SECONDARY OUTCOMES:
Safety and radiation dosimetry of PET tracer [11C] MePPEP; Distribution and variance of CB1 receptors in the brain of healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Carson RE, Huang SC, Green MV. Weighted integration method for local cerebral blood flow measurements with positron emission tomography. J Cereb Blood Flow Metab. 1986 Apr;6(2):245-58. doi: 10.1038/jcbfm.1986.38. PMID 3485644